CLINICAL TRIAL: NCT02556879
Title: Immunization Anti HLA in the Liver Transplant Recipients (DSATH)
Acronym: DSATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P140315
Record Dates: First submitted 2015-08-03; First posted 2015-09-22 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplantation; Graft Failure
Keywords: Liver transplantation; Graft failure; Donor specific antibodies
MeSH Terms: interventions — Gene Library

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liver retransplantation (Other): * Donor specific antibodies :Additional samples for Donor specific at each visit
  * Serum bank : Additional samples for serum bank at each visit if possible
  * DNA banq : Additional sample for DNA banq at inclusion visit if possible
  * Liver biopsy :Liver biopsy at 12 and 24 months after retransplantation (dependind the centers : procedure performed in routine or interventional procedure)
  * Liver ultrasounds and Fibroscan : Liver ultrasounds and Fibroscan at 12 and 24 months after retransplantation (dependind the centers : procedure performed in routine or interventional procedure)
  Interventions: Biological: Donor specific antibodies; Biological: Serum bank; Biological: DNA bank; Procedure: Liver biopsy; Procedure: Liver ultrasounds and Fibroscan

INTERVENTIONS:
Biological: Donor specific antibodies — Additional samples for Donor specific antibodies at each visit
Biological: Serum bank — Additional samples for serum bank at each visit if possible
Biological: DNA bank — Additional sample for DNA bank at inclusion visit if possible
Procedure: Liver biopsy — Liver biopsy at 12 and 24 months after retransplantation (depending the centers : procedure performed in routine or interventional procedure)
Procedure: Liver ultrasounds and Fibroscan — Liver ultrasounds and Fibroscan at 12 and 24 months after retransplantation (depending the centers : procedure performed in routine or interventional procedure)

SUMMARY:
Anti HLA alloimmunization against the donor evaluated by the detection of anti-donor specific antibodies (DSA) is an underestimated factor in liver transplantation and may contribute to dysfunction and graft loss , especially among candidates for retransplantation, that have major immunization.

This study will analyzed immunization markers at the time of liver retransplantation and systematically in patients follow-up. This will allow to characterize the histological lesions due to humoral immunization, to establish further investigations and to adapt early immunosuppressive therapy.

DETAILED DESCRIPTION:
Humoral rejection, related to immunization of the patient against the graft, is diagnosed by the presence of DSA. This serious complication, responsible for dysfunction and graft loss in kidney and heart transplant, is treated by strengthening the immunosuppressive treatment. Humoral rejection is poorly characterized in liver transplantation, but might explain the severe dysfunctions and misunderstood losses of liver transplant. In a preliminary study after liver transplantation, it was observed that the presence of DSAs was more common among patients with unexplained dysfunction (n = 22) compared to patients without dysfunction (n = 69) (95% versus 51%). After liver transplantation, 20% of patients are immunized, against 50% after retransplantation, and after retransplantation, approximately 40% of patients present with graft dysfunction within 2 years.

The role of humoral rejection in graft lesion and loss is unknown after liver transplantation because DSAs are not evaluated and histological lesions associated with DSAs are not analyzed. It is essential to characterize the humoral rejection in liver transplantation or after liver retransplantation (highly immunized population) and immunization markers that are responsible, for early management of this complication by an increased immunosuppressive therapy as it is done for kidney and heart transplantation. This could limit the progression to graft loss.

A specific anti HLA immunization against the donor (DSA - Donor Specific Antibodies) is an underestimated factor in liver transplantation and may contribute to dysfunction and loss of liver graft, especially among candidates for retransplantation, stronger immune.

This study will look for these markers of immunization at the time of liver retransplantation and systematically in patients follow-up. This will allow to characterize the histological lesions, to establish further investigations and to adapt early immunosuppressive therapy.

Methodology, experimental design: prospective, multicenter study. Results of anti HLA antibodies and DSA will not be given not to influence the teams on patient treatment.

Inclusion in the pre-retransplantation visit : obtaining of the informed consent, HLA and anti-HLA antibodies, HLA Typing.

Visit before-ReTH: HLA antibodies and DSA Visit 1 (day of transplant): Standard biology, HLA antibodies and DSA, Crossmatch, Histological analysis of liver de-transplantation locally and centralized.

Visits 2 and 3 (months 1 and 3 post retransplantation) : Standard biology, anti-HLA antibodies and DSA, liver Doppler Ultrasound (as usual the center).

Visits 4 and 5 (months 12 and 24 post retransplantation), and in case of unexplained hepatic dysfunction: Standard biology, HLA antibodies and DSA, liver Doppler-Ultrasound, Fibroscan and hepatic puncture biopsy : histological analysis on site and centralized.

Number of subjects required: 100 patients to be included (200 patients eligible to be selected in pre-transplant consultation for 100 patients retransplanted to include).

Total study duration: up to 6 years (3 years for inclusion and 3 years of follow-up - up to 1 year pre waiting Reth and 2 years post-transplant) Inclusion period: 2 years Duration of participation for a patient: up to 3 years (1 year maximum pre retransplantation waiting + 2 years after transplantation)

Number of participating centers: 11

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with no upper age limit,
* Candidate for a liver retransplantation, whatever the indication, the period or the number of retransplantation
* Recipient of a social protection scheme or entitled
* Signature of informed consent

Exclusion Criteria:

* HIV positive patient,
* Multi-organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Risk of graft failure at 24 months (Odds Ratio) depending on the presence of DSA at retransplantation. | 24 months after retransplantation
  The graft failure is defined by abnormal hepatic tests (AST, ALT, GGT, PAL, total and conjugated bilirubin, PT, INR), and/or abnormal hepatic histology , and/or abnormal hepatic imagery.

SECONDARY OUTCOMES:
Evaluate the association between the presence of the DSA at retransplantation and histological abnormalities of the explant and graft. ( Pearson's chi-square test or Fischer exact test). | retransplantation, 12 and 24 months after retransplantation
  The DSA will be detected by a luminex technology and the positivity will be mesurated by the mean fluorescence intensity. Histological findings of the explant associated with anti HLA immunization will be described and clustered by the approach proposed by Lefaucheur et al (34), the analysis of C4d is conducted.
  The histological abnormalities graft will be evaluated from biopsies performed at 12 and 24 months.
Evaluate the association between the presence of the DSA at before retransplantation and biological abnormalities graft from the previous donor | 9 months, 6 months, 3 months Before transplantation
Evaluate the association between the presence of the DSA at retransplantation and biological abnormalities graft at 1, 3, 12 and 24 months.( Pearson's chi-square test or Fischer exact test). | 1, 3, 12 and 24 months after retransplantation
  The presence of abnormality will be determined from the AST, ALT, GGT, PAL, total and conjugated bilirubin, PT, INR.
Evaluate the association between the presence of DSA and fibrosis Fibroscan measured at 12 and 24 months. (Student t-test or non parametric test). | 12 and 24 months after retransplantation
Evaluate the association between the number of acute rejection episodes and the presence of the DSA at retransplantation and their evolution (especially of recurrence).(Pearson's chi-square test or Fischer exact test). | 24 months after retransplantation

CONTACTS AND LOCATIONS:
Overall Officials: PERDIGAO Fabiano, PH, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Unité Médicale de Transplantation Hépatique In Service d'Hépato-Gastro-Entérologie, Päris, France